CLINICAL TRIAL: NCT02792166
Title: Single Anastomosis Duodeno-ileal Bypass With Sleeve Gastrectomy (SADI-S): A Prospective Cohort Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Amin Andalib, MD MSc FRCSC, McGill University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-588 MUHC
Record Dates: First submitted 2016-06-02; First posted 2016-06-07 (Estimated); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Obesity; Morbid Obesity
Keywords: Morbid obesity; Metabolic syndrome; Metabolic surgery; Bariatric surgery; SADI; BPD-DS
MeSH Terms: conditions — Obesity; Obesity, Morbid; Metabolic Syndrome | interventions — Bariatric Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BPD-DS (Active Comparator): BPD-DS involves creating a sleeve gastrectomy and creation of a Roux-en-Y bypass involving a Roux limb (150cm) which is anastomosed to the transected first-stage of the duodenum and a short common channel (100cm).
  Interventions: Procedure: BPD-DS
- SADI-S (Experimental): SADI-S involves creating a sleeve gastrectomy but simplifies the bypass part of the BPD-DS by a single anastomosis of a loop of jejunum at 250cm from the ileocecal valve (longer common channel) to the transected first-stage of the duodenum instead of the Roux-en-Y construct.
  Interventions: Procedure: SADI-S

INTERVENTIONS:
Procedure: BPD-DS — Biliopancreatic Diversion with Duodenal Switch
  Other Names: Bariatric/metabolic surgery
  Arms: BPD-DS
Procedure: SADI-S — Single Anastomosis Duodeno-ileal Bypass with Sleeve Gastrectomy
  Other Names: Bariatric/metabolic surgery
  Arms: SADI-S

SUMMARY:
The prevalence of morbid obesity in Canada has risen almost 5 fold in the past three decades. Surgery remains the cornerstone of treatment of obesity and related comorbidities such as type-2 diabetes. Bariatric/metabolic procedures can be classified into 2 main categories: a) those that cause restriction, and b) those that add a malabsorptive component to restriction. Currently sleeve gastrectomy (SG), which is a purely restrictive operation, is the most frequently performed procedure in North America.

Interestingly, combined restrictive/malabsorptive procedures such as Roux-en-Y gastric bypass (RYGB) or biliopancreatic diversion with duodenal switch (BPD-DS) are more effective procedures when compared to purely restrictive ones. Moreover, the conventional BPD-DS procedure has been shown to be significantly more effective than RYGB in achieving durable weight loss and resolving comorbidities such as type-2 diabetes. Despite superior outcomes, the performance of BPD-DS is highly institution dependant and comprises less than 5% of the annual bariatric procedures performed worldwide.

Common reservations against BPD-DS are related to the side effects of the procedure, and include frequent bowel movements, flatulence, fat, micronutrient and protein malnutrition. Furthermore, longer operative times and surgical technical challenges are also reasons for lower prevalence of the BPD-DS procedure.

Single anastomosis duodeno-ileal bypass with sleeve gastrectomy (SADI-S) is a modification of the conventional BPD-DS that potentially addresses many of these concerns. In addition, it is a suitable second-stage or salvage procedure for severely obese patients with inadequate weight loss or resolution of obesity-related comorbidities after SG. Despite showing excellent results of up to 5 years with acceptable postoperative morbidity, all the literature on SADI-S originates from a single center and has not been compared directly with BPD-DS. Hence, the investigators aim to evaluate the feasibility, safety, and postoperative outcomes of SADI-S as it compares to conventional BPD-DS in morbidly obese patients.

This project has three specific aims:

1. To evaluate feasibility and short-term safety of SADI-S.
2. To evaluate short and long-term beneficial outcomes.
3. To evaluate and compare long-term morbidity.

DETAILED DESCRIPTION:
The prevalence of morbid obesity in Canada has risen almost 5 fold in the past three decades. Surgery remains the cornerstone of treatment of obesity and related comorbidities such as type-2 diabetes. Bariatric/metabolic procedures can be classified into 2 main categories: a) those that cause restriction, and b) those that add a malabsorptive component to restriction. Currently sleeve gastrectomy (SG), which is a purely restrictive operation, is the most frequently performed procedure in North America.

Interestingly, combined restrictive/malabsorptive procedures such as Roux-en-Y gastric bypass (RYGB) or biliopancreatic diversion with duodenal switch (BPD-DS) are more effective procedures when compared to purely restrictive ones. Moreover, the conventional BPD-DS procedure has been shown to be significantly more effective than RYGB in achieving durable weight loss and resolving comorbidities such as type-2 diabetes. Despite superior outcomes, the performance of BPD-DS is highly institution dependant and comprises less than 5% of the annual bariatric procedures performed worldwide.

Common reservations against BPD-DS are related to the side effects of the procedure, and include frequent bowel movements, flatulence, fat, micronutrient and protein malnutrition. Furthermore, longer operative times and surgical technical challenges are also reasons for lower prevalence of the BPD-DS procedure.

Single anastomosis duodeno-ileal bypass with sleeve gastrectomy (SADI-S) is a modification of the conventional BPD-DS that potentially addresses many of these concerns. In addition, it is a suitable second-stage or salvage procedure for severely obese patients with inadequate weight loss or resolution of obesity-related comorbidities after SG. Despite showing excellent results of up to 5 years with acceptable postoperative morbidity, all the literature on SADI-S originates from a single center and has not been compared directly with BPD-DS. Hence, the investigators aim to evaluate the feasibility, safety, and postoperative outcomes of SADI-S as it compares to conventional BPD-DS in morbidly obese patients. Our project has three specific aims:

1. To evaluate feasibility and short-term safety of SADI-S. The investigators will assess operative parameters (e.g. procedure time, inadvertent injuries, need for conversion to laparotomy, and transfusion of blood products) and 30-day postoperative adverse events (e.g. length of stay, superficial/deep surgical site infection, leak, venous thromboembolism (VTE), need for reintervention and readmission).
2. To evaluate short and long-term beneficial outcomes. The investigators will evaluate and compare excess weight loss, resolution of type-2 diabetes and other comorbidities, and changes in quality of life at 1, 6, 12 months and yearly thereafter for both groups.
3. To evaluate and compare long-term morbidity. The investigators will evaluate and compare both groups at 6, 12 months and yearly thereafter following surgery for long-term morbidities (e.g. frequency of bowel movements, fat malabsorption, micronutrient and protein-calorie malnutrition, need for supplemental nutrition, internal/incisional hernia, and gastro-esophageal reflux).

ELIGIBILITY:
Inclusion Criteria:

Participants must meet ALL of the following inclusion criteria:

* Age ≥18 years and ≤60 years
* Fulfill criteria for bariatric surgery as coined by National Institutes of Health
* Give written informed consent

Exclusion Criteria:

Participants who meet any of the following criteria at the time of the baseline visit are excluded from the study:

* Presence of the following baseline comorbidities:
* Congestive heart failure (CHF),
* Chronic kidney disease (CKD) stage 3-5 (or GFR <60 ml/min per 1.73 m2),
* Inflammatory bowel disease (IBD),
* Pulmonary hypertension (PHTN),
* Cirrhosis.
* Severe gastroesophageal reflux disorder (GERD) +/- presence of any Barrett's disease
* Individuals who were found by any member of the multidisciplinary team (nutritionist, nurse, psychologist, and surgeon) to be at risk for lack of support and poor compliance (e.g. ≥2 missed appointments without a valid justification)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2016-06; Primary Completion 2019-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Short-term Safety Assessment | 30 days
  To evaluate feasibility and short-term safety of SADI-S, we will assess operative parameters (procedure time, inadvertent injuries, need for conversion to laparotomy, and transfusion of blood products) and 30-day postoperative adverse events (length of stay, superficial/deep surgical site infection, leak, venous thromboembolism (VTE), need for reintervention and readmission).
Weight loss | 5 years
  %EWL and change in BMI as compared to preoperative reference values

SECONDARY OUTCOMES:
Long-term Morbidity Assessment | 5 years
  Postoperatively at 1, 6, 12 months and yearly thereafter for 5 years both groups will be compared for incidence of long-term morbidities including frequency of bowel movements, fat malabsorption, micronutrient and protein-calorie malnutrition, need for supplemental nutrition, internal/incisional herniation, and worsening versus de novo GERD.
  At each visit protein (albumin, total protein) and vitamin/micronutrient levels (calcium, magnesium, iron, zinc, copper, selenium, vitamins A/E/D/K/B1/B6/B12) will be monitored using respective blood tests.
Remission of T2DM | 5 years
  The presence of T2DM will be diagnosed according to the American Diabetes Association's current criteria:
  1. HbA1C ≥6.5 percent, OR
  2. FPG ≥126 mg/dL (7.0 mmol/L), OR
  3. 2-hour plasma glucose ≥200 mg/dL (11.1 mmol/L) during an OGTT, OR
  4. In a patient with classic symptoms of hyperglycemia or hyperglycemic crisis, a random plasma glucose ≥200 mg/dL (11.1 mmol/L)
Resolution/Improvement in other obesity related comorbidities | 5 years
  Hypertension, Dyslipidemia, Obstructive sleep apnea, NAFLD/NASH
Quality of Life Assessment | 5 years
  Quality of life status will be assessed using the SF-36 questionnaire at each follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Amin Andalib, MD MSc FRCSC, Principal Investigator — McGill University
Locations (1):
- McGill University Health Center, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sanchez-Pernaute A, Herrera MA, Perez-Aguirre ME, Talavera P, Cabrerizo L, Matia P, Diez-Valladares L, Barabash A, Martin-Antona E, Garcia-Botella A, Garcia-Almenta EM, Torres A. Single anastomosis duodeno-ileal bypass with sleeve gastrectomy (SADI-S). One to three-year follow-up. Obes Surg. 2010 Dec;20(12):1720-6. doi: 10.1007/s11695-010-0247-3. PMID 20798995
- [Result] Sanchez-Pernaute A, Rubio MA, Cabrerizo L, Ramos-Levi A, Perez-Aguirre E, Torres A. Single-anastomosis duodenoileal bypass with sleeve gastrectomy (SADI-S) for obese diabetic patients. Surg Obes Relat Dis. 2015 Sep-Oct;11(5):1092-8. doi: 10.1016/j.soard.2015.01.024. Epub 2015 Feb 7. PMID 26048517
- [Result] Sanchez-Pernaute A, Rubio MA, Perez Aguirre E, Barabash A, Cabrerizo L, Torres A. Single-anastomosis duodenoileal bypass with sleeve gastrectomy: metabolic improvement and weight loss in first 100 patients. Surg Obes Relat Dis. 2013 Sep-Oct;9(5):731-5. doi: 10.1016/j.soard.2012.07.018. Epub 2012 Aug 7. PMID 22963820
- [Result] Sanchez-Pernaute A, Rubio MA, Conde M, Arrue E, Perez-Aguirre E, Torres A. Single-anastomosis duodenoileal bypass as a second step after sleeve gastrectomy. Surg Obes Relat Dis. 2015 Mar-Apr;11(2):351-5. doi: 10.1016/j.soard.2014.06.016. Epub 2014 Jul 10. PMID 25543309
- [Result] Sanchez-Pernaute A, Rubio Herrera MA, Perez-Aguirre E, Garcia Perez JC, Cabrerizo L, Diez Valladares L, Fernandez C, Talavera P, Torres A. Proximal duodenal-ileal end-to-side bypass with sleeve gastrectomy: proposed technique. Obes Surg. 2007 Dec;17(12):1614-8. doi: 10.1007/s11695-007-9287-8. Epub 2007 Nov 27. PMID 18040751
- [Derived] Andalib A, Safar A, Bouchard P, Demyttenaere S, Court O. Single Anastomosis Duodenal Switch versus Classic Duodenal Switch: Long-term Outcomes from a Prospective Comparative Cohort Study. Obes Surg. 2023 Dec;33(12):3951-3961. doi: 10.1007/s11695-023-06900-z. Epub 2023 Oct 21. PMID 37864735
- [Derived] Andalib A, Bouchard P, Alamri H, Bougie A, Demyttenaere S, Court O. Single anastomosis duodeno-ileal bypass with sleeve gastrectomy (SADI-S): short-term outcomes from a prospective cohort study. Surg Obes Relat Dis. 2021 Feb;17(2):414-424. doi: 10.1016/j.soard.2020.09.015. Epub 2020 Sep 14. PMID 33158766